CLINICAL TRIAL: NCT02005965
Title: The Low Rectal Cancer Study.
Brief Title: Low Rectal Cancer Study (MERCURY II)
Acronym: MERCURY II
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CCR2943
Record Dates: First submitted 2013-11-21; First posted 2013-12-09 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Adenocarcinoma; Adenocarcinoma, Mucinous; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Cystic, Mucinous, and Serous; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases
Keywords: Rectal Cancer; Low Rectal Cancer; MERCURY; Cancer; CRM; Circumferential Margin; Quality of Life; MRI; Radiology; Abdominoperineal Excision; Anterior Resection; Surgery; Pathology
MeSH Terms: conditions — Adenocarcinoma; Adenocarcinoma, Mucinous; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Cystic, Mucinous, and Serous; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Staging and outcomes for patients with Low Rectal Cancer: Low Rectal Cancer defined on MRI as a cancer within 6cm of the anal verge

SUMMARY:
The MERCURY Study demonstrated the accuracy, feasibility and reproducibility of Magnetic Resonance Imaging (MRI) to stage rectal cancer in a prospective, multidisciplinary, multi-centre study. However, there were differences in patient outcome, dependent upon the position of the tumour in the rectum and its height above the anal verge. Whilst the outcome was excellent for patients who underwent an anterior resection, the outcome, based upon margin involvement and quality of the specimen, was poor for patients who underwent an abdomino-perineal excision for low rectal cancer.

It is proposed that accurate MRI staging pre-operatively will allow the correct patients to receive neo-adjuvant chemoradiotherapy (CRT), and also pre-warn the surgeons if the resection margins appear threatened so that the operation can be modified to take this into account. The primary aims of the Low Rectal Cancer Study (MERCURY II) are to assess the rate of CRM positivity rate in low rectal cancer and to assess the difference in global quality of life at two years post surgery in patients according to plane of surgery with or without sphincter preservation.

DETAILED DESCRIPTION:
The aim of this study is to reduce the positive margin rate of 30% to around 15%. The study is an international multicentre, prospective, observational study, whereby patients with biopsy-proven low-rectal cancer (lower edge of the tumour < 6cms from the anal verge on MRI), will be recruited from participating centres, having given informed, written consent. Data from the radiology, surgical and pathological aspects will be collected and analysed centrally at the Royal Marsden Hospital. The patient's medical records will be reviewed for five years post surgery, and the patients will also be followed up by quality of life questionnaires. This project aims to show that in low rectal cancer, improved local control and survival can be achieved through a reduction in the involved CRM rates by MRI-planned surgery and selective pre-operative therapy. It also aims to assess the ability to predict disease recurrence and to provide an assessment of disease-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed, written consent.
* Adults age 18 or over - male or female.
* Recently diagnosed with biopsy-proven, primary, low rectal cancer.
* No previous therapy for rectal cancer.

Exclusion Criteria:

* Current pregnancy, including ectopic pregnancy.
* Previous pelvic/rectal malignancy (excluding carcinoma in-situ).
* Previous pelvic radiotherapy.
* Previous pelvic floor surgery for faecal incontinence or prolapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven adenocarcinoma within 6cm of the anal verge confirmed on MRI.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2007-08-13 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2021-03-11 (Estimated)

PRIMARY OUTCOMES:
To assess the rate of CRM positivity rate in low rectal cancer. | 4 years
To compare global quality of life at two years post surgery in patients according to plane of surgery with or without sphincter preservation. | 8 years

SECONDARY OUTCOMES:
To compare patient reported outcomes in patients according to plane of surgery with or without sphincter preservation. | 8 years
Analysis of the clinical and radiological factors influencing the decision by surgeons to carry out Anterior Resections, APE or extralevator APE. | 8 years
Comparison of time to local recurrence, disease-free and overall survival between patients undergoing different types of surgery. | 8 years
Comparison of imaging and pathology staging assessment, patient characteristics and complication rates, between different types of surgery and surgical approaches. | 8 years
Investigation of potential associations between imaging and pathology assessment of radial and distal margins, neo-adjuvant chemoradiotherapy, perineal complications and sphincter preservation rates. | 8 years
Investigation of potential association between length of operation with number of complications and length of post-operative ITU/HDU stay. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, Principal Investigator — Royal Marsden NHS Foundation Trust; Brendan Moran, Principal Investigator — Pelican Cancer Foundation
Locations (17):
- Germany (2):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Krankenhaus Dresden-Friedrichstadt, Dresden
- The First Surgical Clinic, Belgrade, Serbia
- United Kingdom (14):
  - Milton Keynes General Hospital, Milton Keynes, Buckinghamshire
  - Stepping Hill Hospital, Stockport, Cheshire
  - North Hampshire Hospitals NHS Trust (Basingstoke Hospital), Basingstoke, Hampshire
  - West Middlesex University Hospital, Isleworth, Middlesex
  - Weston General Hospital, Weston-super-Mare, Somerset
  - Croydon University Hospital, Croydon, Surrey
  - Frimley Park Hospital NHS Foundation Trust, Frimley, Surrey
  - Princess of Wales Hospital, Bridgend, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Salisbury NHS Foundation Trust (Salisbury District Hospital), Salisbury, Wiltshire
  - Ulster Hospital, Belfast
  - Royal Marsden Hospital, London & Surrey
  - North Manchester General Hospital, Manchester

REFERENCES:
- [Derived] Battersby NJ, How P, Moran B, Stelzner S, West NP, Branagan G, Strassburg J, Quirke P, Tekkis P, Pedersen BG, Gudgeon M, Heald B, Brown G; MERCURY II Study Group. Prospective Validation of a Low Rectal Cancer Magnetic Resonance Imaging Staging System and Development of a Local Recurrence Risk Stratification Model: The MERCURY II Study. Ann Surg. 2016 Apr;263(4):751-60. doi: 10.1097/SLA.0000000000001193. PMID 25822672